CLINICAL TRIAL: NCT01918358
Title: A Randomized, Open-label, Single Dose Crossover Study to Compare the Safety and Pharmacokinetics Between Fixed-dose Combination VR 160/20 mg and Co-administration of Diovan® (Valsartan) Film-coated Tablet 160 mg and Crestor® (Rosuvastatin) 20 mg in Healthy Male Volunteers
Brief Title: Safety and Pharmacokinetics Between Fixed-dose Combination VR 160/20 mg and Co-administration of Diovan® (Valsartan) Film-coated Tablet 160 mg and Crestor® (Rosuvastatin) 20 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-VRCL005
Record Dates: First submitted 2013-08-05; First posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Valsartan; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fixed-dose combination VR 160/20 mg-1 (Experimental): Fixed-dose combination VR 160/20 mg-1 is administered by mouth at Day 1, 8 and 15.
  Interventions: Drug: Sequence 1 : Period 1 (VR 160/20 mg-1), Period 2(VR 160/20 mg-2), Period (V+R); Drug: Sequence 2 : Period 1 (VR 160/20 mg-2), Period 2 (V+R), Period 3 (VR 160/20 mg-1); Drug: Sequence 3 : Period 1 (V+R), Period 2 (VR 160/20 mg-2), Period 3 (VR 160/20 mg-1); Drug: Sequence 4 : Period 1 (VR 160/20 mg-1), Period 2 (V+R), Period 3 (VR 160/20 mg-2 ); Drug: Sequence 5 : Period 1 (VR 160/20 mg-2), Period 2 (VR 160/20 mg-1), Period 3 (V+R ); Drug: Sequence 6 : Period 1 (V+R), Period 2 (VR 160/20 mg-1), Period 3 (VR 160/20 mg-2)
- Fixed-dose combination VR 160/20 mg-2 (Experimental): Fixed-dose combination VR 160/20 mg-2 is administered by mouth at Day 1, 8 and 15.
  Interventions: Drug: Sequence 1 : Period 1 (VR 160/20 mg-1), Period 2(VR 160/20 mg-2), Period (V+R); Drug: Sequence 2 : Period 1 (VR 160/20 mg-2), Period 2 (V+R), Period 3 (VR 160/20 mg-1); Drug: Sequence 3 : Period 1 (V+R), Period 2 (VR 160/20 mg-2), Period 3 (VR 160/20 mg-1); Drug: Sequence 4 : Period 1 (VR 160/20 mg-1), Period 2 (V+R), Period 3 (VR 160/20 mg-2 ); Drug: Sequence 5 : Period 1 (VR 160/20 mg-2), Period 2 (VR 160/20 mg-1), Period 3 (V+R ); Drug: Sequence 6 : Period 1 (V+R), Period 2 (VR 160/20 mg-1), Period 3 (VR 160/20 mg-2)
- Valsartan 160mg placebo + Rosuvastatin 20mg (Experimental): Both Valsartan 160mg placebo and Rosuvastatin 20mg are administered by mouth at Day 1, 8 and 15.
  Interventions: Drug: Sequence 1 : Period 1 (VR 160/20 mg-1), Period 2(VR 160/20 mg-2), Period (V+R); Drug: Sequence 2 : Period 1 (VR 160/20 mg-2), Period 2 (V+R), Period 3 (VR 160/20 mg-1); Drug: Sequence 3 : Period 1 (V+R), Period 2 (VR 160/20 mg-2), Period 3 (VR 160/20 mg-1); Drug: Sequence 4 : Period 1 (VR 160/20 mg-1), Period 2 (V+R), Period 3 (VR 160/20 mg-2 ); Drug: Sequence 5 : Period 1 (VR 160/20 mg-2), Period 2 (VR 160/20 mg-1), Period 3 (V+R ); Drug: Sequence 6 : Period 1 (V+R), Period 2 (VR 160/20 mg-1), Period 3 (VR 160/20 mg-2)

INTERVENTIONS:
Drug: Sequence 1 : Period 1 (VR 160/20 mg-1), Period 2(VR 160/20 mg-2), Period (V+R)
  Other Names: Rovatitan tab; Diovan; Crestor
Drug: Sequence 2 : Period 1 (VR 160/20 mg-2), Period 2 (V+R), Period 3 (VR 160/20 mg-1)
  Other Names: Rovatitan tab; Diovan; Crestor
Drug: Sequence 3 : Period 1 (V+R), Period 2 (VR 160/20 mg-2), Period 3 (VR 160/20 mg-1)
  Other Names: Rovatitan tab; Diovan; Crestor
Drug: Sequence 4 : Period 1 (VR 160/20 mg-1), Period 2 (V+R), Period 3 (VR 160/20 mg-2 )
  Other Names: Rovatitan tab; Diovan; Crestor
Drug: Sequence 5 : Period 1 (VR 160/20 mg-2), Period 2 (VR 160/20 mg-1), Period 3 (V+R )
  Other Names: Rovatitan tab; Diovan; Crestor
Drug: Sequence 6 : Period 1 (V+R), Period 2 (VR 160/20 mg-1), Period 3 (VR 160/20 mg-2)
  Other Names: Rovatitan tab; Diovan; Crestor

SUMMARY:
To compare the safety and pharmacokinetics between ROVATITAN tab. 160/20 mg (ROVATITAN tab 160/20mg-1, ROVATITAN tab. 160/20mg-2) and coadministration of Diovan® (Valsartan) 160 mg and Crestor® (Rosuvastatin) 20 mg in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male aged 20~45 years at screening
2. 19 kg/m2 ≤ BMI ≤27 kg/m2 at screening
3. Subject who is able to communicate with investigators and understand the nature of the clinical study and is willing and able to provide a written informed consent form

Exclusion Criteria:

1. Subject with current or previous clinically significant diseases in liver, renal, neurologic, pulmonary, gastrointestinal, endocrine, hematologic, oncologic, cardiovascular, psychological, and musculoskeletal system
2. Patient with renal defects (Calculated GFR < 60 ml/min based on serum creatinine level )
3. Subject who can not satisfy the following criteria for sitting blood pressure at screening test 90 ≤SBP <140 (mmHg) 60 ≤ DBP <90 (mmHg)
4. Subject who can not satisfy the following criteria at screening 1) AST and ALT ≤ 1.5x ULN 2) Serum total bilirubin ≤ 1.5x ULN 3) CK (Creatinine kinase) ≤ 2x ULN
5. Subject with a medical history of gastrointestinal diseases (e.g., Crohn's disease, ulcer) or a surgery (for appendicitis and hernia repair are allowed) that might affect the investigational product absorption
6. Subject with hypersensitivity to the drugs containing components of valsartan and rosuvastatin or other drugs (aspirin, antibiotics) or a previous clinically significant history of hypersensitivity
7. Subject with a previous history of drug overdose or a positive to the drugs (Barbiturate, Benzodiazepine, Methamphetamine, Cannabinoids, Cocaine, Opiate) in urine drug screening test
8. Subject who has taken any prescribed medicines or oriental medicines within two weeks before the first investigational product administration, or who has taken any over-the-counter drugs within one week before the first investigational product administration (If the subject is eligible for all other criteria, he or she may participate in the clinical study based on investigator's discretion.)
9. Subject who has taken other investigational products within 60 days before the first investigational product administration
10. Subject who donated whole blood within 60 days or donated apheresis blood within 30 days or received a transfusion within 30 days before the first investigational product administaration.
11. Subject who has taken the drugs that induce or inhibit drug-metabolizing enzymes such as barbiturates within 30 days before the first investigational product administration
12. Subject with a daily intake of drinks containing caffeine (coffee, tea, coke) or grapefruit juice > average of 4 cups / day (800 mL) or a subject who can not discontinue such drinks during the clinical study period(from screening to post-study visit)
13. Subject with a mean weekly drinking amount of > 140g or a subject who can not stop drinking until outpatient visit after the investigational product administration, including the hospitalization in each period.
14. Subject with a mean daily smoking amount of > 10 cigarettes or a subject who can not stop smoking during the hospitalization
15. Subject positive result in serology tests (hepatitis B, hepatitis C, HIV)
16. Subject with genetic muscle disease, or familial history of muscle disease, or medical history of drug-derived muscle disorder
17. Subject who is considered not to be eligible at investigator's discretion.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Cmax of valsartan and rosuvastatin | 0h(pre-dosing), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 6h, 8h, 12h, 24h, 48h for each period (total 16 times)
AUC last of valsartan and rosuvastatin | 0h(pre-dosing), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 6h, 8h, 12h, 24h, 48h for each period (total 16 times)

OTHER OUTCOMES:
Safety evaluation | -28~-2d, 1d, 2d, 3d, 8d, 9d, 10d, 15d, 16d, 17d, 21 ± 2d
  The severity of adverse events and their relationship with the investigational products are schematized by treatment group. Descriptive statistics are calculated for the frequency, percentage, 12-lead ECG and clinical laboratory tests results of the subjects who have adverse events and the results of each item are reviewed.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea